CLINICAL TRIAL: NCT04930211
Title: The Effectiveness of Lumbar Transforaminal Anterior Epidural Steroid Injections in Discogenic Low Back Pain Associated With Modic Type-1 Change
Brief Title: Lumbar Transforaminal Anterior Epidural Steroid Injections in Discogenic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.2020.961
Record Dates: First submitted 2021-05-01; First posted 2021-06-18 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Degenerative Disc Disease; Low Back Pain
Keywords: transforaminal epidural injection; degenerative disc disease; modic changes
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modic Type-1 changes (Active Comparator): Transforaminal Epidural Steroid Injection will be performed on patients at the pathology detected level bilaterally. The Kambin approach will be preferred in order to reach the intervertebral disc.
  Interventions: Drug: Dexamethasone-Lidocaine
- Degenerative disc disease without Modic Type-1 changes (Active Comparator): Transforaminal Epidural Steroid Injection will be performed on patients at the pathology detected level bilaterally. The Kambin approach will be preferred in order to reach the intervertebral disc.
  Interventions: Drug: Dexamethasone-Lidocaine

INTERVENTIONS:
Drug: Dexamethasone-Lidocaine — Kambin's triangle approach in transforaminal epidural injection: Kambin's triangle is defined as a right triangle over the dorsolateral disc. The hypotenuse is the exiting nerve root, the base is the superior border of the caudal vertebra, and the height is the dura/traversing nerve root. it is possible to inject agents at the entrance and middle zone as the main areas of nerve entrapment by injecting at the retrodiscal area of the entrance zone, as proximal area of the targeted nerve root.
  Other Names: Transforaminal epidural steroid injection

SUMMARY:
Modic changes have been associated with low back pain in many clinical studies and are often considered a part of the disc degeneration process. Modic type 1 change is considered an inflammatory process. The aim of this study is to determine the effectiveness of lumbar transforaminal epidural steroid injections in Modic type-1 changes.

DETAILED DESCRIPTION:
Modic changes have been associated with low back pain in many clinical studies and are often considered a part of the disc degeneration process. However, in degenerative disc disease, whether the pain could be attributed to Modic changes or not is still a matter of debate.

There are different options in the treatment of low back pain due to degenerative disc disease (DDD) and Modic changes. Conservative treatments and surgical approaches are some of them. Other interventional procedures include intradiscal and epidural steroid injections which have relatively less risk of complications than surgery.

The only study in the literature investigating the effectiveness of epidural steroid injections in patients with low back pain associated with modic changes belongs to Butterman et al. They reported that patients with Modic changes (type 1) responded better to epidural steroid injections than those without endplate irregularities. However, they did not report the details of the procedure, such as the steroid and local anesthetic they used, the amount of them and the level of the procedure. Moreover, they used different approaches including interlaminar and transforaminal, which may be misleading while interpreting the results.

Based on these results, the aim of this study is to determine the effectiveness of lumbar transforaminal epidural steroid injections in Modic type-1 changes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Non-radicular, axial back pain
* Lack of response to conservative treatments
* Detection of Modic type 1 changes in contrast-enhanced Lumbar MRI or intervertebral disc findings that may be associated with discogenic pain (nuclear signal intensity change in the disc [black disc], height loss, or high-intensity zone)

Exclusion Criteria:

* Patients younger than 18 and older than 65
* Describing pain radiating to the lower extremity (those with radicular pain)
* Nerve root compression due to disc herniation or other reasons
* Modic changes in more than one level
* Positive facet loading test
* Spinal stenosis or spondylolisthesis
* Diagnosed with spondylodiscitis
* Pregnancy
* Patients with inflammatory rheumatic diseases
* Patients whose use of non-steroidal anti-inflammatory drugs is contraindicated (renal failure, bleeding disorders, etc.)
* Patients with exercise intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-05 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale | Baseline
  a scale used to measure the severity of pain. "0" is scored as no pain, "10" as the most severe pain that could be. The patient scores between 0 and 10 for pain.
numeric rating scale | first month
  a scale used to measure the severity of pain. "0" is scored as no pain, "10" as the most
numeric rating scale | third month
  a scale used to measure the severity of pain. "0" is scored as no pain, "10" as the most
numeric rating scale | sixth month
  a scale used to measure the severity of pain. "0" is scored as no pain, "10" as the most

SECONDARY OUTCOMES:
Oswestry disability index | Baseline
  a functional disability index used in low back pain. The Oswestry Disability Index (ODI) consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. There are six statements under each item, marking what is appropriate for the patient's condition. The first statement is scored as "0" and the sixth statement as "5". The higher the total score, the higher the level of disability.
Oswestry disability index | first month
  a functional disability index used in low back pain. The Oswestry Disability Index (ODI) consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. There are six statements under each item, marking what is appropriate for the patient's condition. The first statement is scored as "0" and the sixth statement as "5". The higher the total score, the higher the level of disability.
Oswestry disability index | third month
  a functional disability index used in low back pain. The Oswestry Disability Index (ODI) consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. There are six statements under each item, marking what is appropriate for the patient's condition. The first statement is scored as "0" and the sixth statement as "5". The higher the total score, the higher the level of disability.
Oswestry disability index | sixth month
  a functional disability index used in low back pain. The Oswestry Disability Index (ODI) consists of 10 items. The items question the severity of pain, self-care, lifting-carrying, walking, sitting, standing, sleep, the degree of pain change, travel and social life. There are six statements under each item, marking what is appropriate for the patient's condition. The first statement is scored as "0" and the sixth statement as "5". The higher the total score, the higher the level of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Kokar, M.D., Principal Investigator — Saniurfa Education and Research Hospital
Locations (1):
- Marmara University, Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjaer P, Korsholm L, Bendix T, Sorensen JS, Leboeuf-Yde C. Modic changes and their associations with clinical findings. Eur Spine J. 2006 Sep;15(9):1312-9. doi: 10.1007/s00586-006-0185-x. Epub 2006 Aug 9. PMID 16896838
- [Background] Jensen RK, Leboeuf-Yde C, Wedderkopp N, Sorensen JS, Jensen TS, Manniche C. Is the development of Modic changes associated with clinical symptoms? A 14-month cohort study with MRI. Eur Spine J. 2012 Nov;21(11):2271-9. doi: 10.1007/s00586-012-2309-9. Epub 2012 Apr 24. PMID 22526703
- [Background] Kallewaard JW, Terheggen MA, Groen GJ, Sluijter ME, Derby R, Kapural L, Mekhail N, van Kleef M. 15. Discogenic low back pain. Pain Pract. 2010 Nov-Dec;10(6):560-79. doi: 10.1111/j.1533-2500.2010.00408.x. Epub 2010 Sep 6. PMID 20825564
- [Background] Buttermann GR. The effect of spinal steroid injections for degenerative disc disease. Spine J. 2004 Sep-Oct;4(5):495-505. doi: 10.1016/j.spinee.2004.03.024. PMID 15363419